CLINICAL TRIAL: NCT03218475
Title: Magnetic Resonance-Guided Focused Ultrasound Combined With Radiotherapy for Palliation of Head and Neck Cancer - A Pilot Study
Brief Title: MRG FU With Radiotherapy for Palliation of H&N Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: On hold pending amendment approval
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Principal Investigator, Dr. Irene Karam, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 229-2016
Record Dates: First submitted 2017-02-16; First posted 2017-07-14 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR Guided Focused Ultrasound (Experimental)
  Interventions: Other: MR Guided Focused Ultrasound

INTERVENTIONS:
Other: MR Guided Focused Ultrasound — Two treatments of focused ultrasound under MRI guidance

SUMMARY:
Head and neck cancer is the sixth most common form of malignancy world-wide. Surgery, chemotherapy and radiation are associated with a high burden of side effects; tumour recurrence within the neck continues to be a major cause of treatment failure. To our knowledge, this research is the first clinical study in human subjects to utilize magnetic resonance guided focused ultrasound to treat cancer of the neck. The goal is to evaluate the safety and technical feasibility of this therapy in order to guide future clinical applications such as ablation, radiosensitization or drug delivery that could ultimately improve clinical outcomes. A total of 10 patients will be treated with MR guided focused ultrasound.

DETAILED DESCRIPTION:
This is a single institution, prospective pilot study to evaluate the safety and feasibility of MR guided focused ultrasound treatment for cancer of the neck in 10 patients. The procedure will consist of a planning MRI scan and two treatment sessions where real time MRI thermometry is used in conjunction with a focused beam to heat the tissue to 40-42oC in the target field over a period of 20-30 seconds per treatment. All patients on the study will undergo palliative radiotherapy and/or chemotherapy. MRg-FU treatments will be delivered on fraction #1 and fraction #10 (50 Gy/20 regimen) or on fraction #1 and fraction #3 (35-45 Gy/5 SBRT regimen). Palliative radiotherapy treatment will be administered to the treatment target lesion and in addition may encompass other tumour regions of the head and neck. The prescribed dose for patients who have not received previous radiotherapy will be between 50Gy over 4 weeks using IMRT or VMAT -based planning or 35-45 Gy in 5 fractions using SBRT technique; in previously irradiated patients, the dose will be determined at the discretion of the treating radiation oncologist. The patient will be assessed by a physician investigator and clinical research assistant (CRA) on the MRg-FU treatment dates, then 1 day, 1 week, 2 weeks, 1 month and 3 months afterward.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to give informed consent
* Weight <140kg
* Biopsy-proven diagnosis of squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma from any primary site with demonstrated metastatic nodal disease in the head and neck region
* Assessed by the treating surgeon, and radiation oncologist, and following a multidisciplinary discussion, determined to have unresectable and/or inoperable disease in the head and neck region in the presence or absence of distant metastases.
* Radiologic evidence of neck lymphadenopathy with at least one target lesion measuring > 1cm in largest dimension. (Recurrent or initial presentation)
* Assessed by the treating radiation/medical oncologists to undergo palliative radiotherapy and/or chemotherapy
* Target lesion visible by non-contrast MRI
* Target lesion accessible for MRg-FU procedure
* Able to communicate sensation during MRg-FU treatment

Exclusion Criteria:

* Pregnant / Nursing woman
* Unable to have contrast-enhanced MRI scan - standard institutional criteria
* Head and neck surgery(excluding biopsy) ≤ 6 weeks prior to study enrolment
* Chemotherapy ≤ 6 weeks prior to enrolment
* Previous radiotherapy to target region ≤ 6 weeks prior to enrolment
* Target lesion involves the skin surface causing ulceration, bleeding or discharge
* Target lesion in contact with hollow viscera
* Target lesion located in skull, spine, or mandible
* Fibrotic scar along proposed HIFU beam path
* Orthopaedic implant along proposed HIFU beam path or at site of target lesion.
* Severe cardiovascular, neurological, renal or hematological chronic disease
* ECOG (Eastern Cooperative Oncology Group) Performance Status ≥ 3.
* Active infection
* Unable to tolerate required stationary position during treatment
* Allergy to MRI contrast agent or sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Toxicity Assessment of MRg-FU Treatment to the Head and Neck Region. | 90 days
  The number, type and severity of adverse effects as assessed using NCI CTCAE v4.03.
Feasibility of MRg-FU Treatments to the Head and Neck Region | 90 days
  The number of patients that meet the eligibility criteria and are able to complete the study treatment protocol.

SECONDARY OUTCOMES:
Treatment Effect | 90 days
  Assessment of changes caused by MR guided FU within the treated tumour region based on post treatment MRI

CONTACTS AND LOCATIONS:
Overall Officials: Irene Karam, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada